CLINICAL TRIAL: NCT02710838
Title: The Feasible Research of Infrared Endoscope to Diagnose Early Gastric Cancer and Evaluate the Invasive Depth of Tumors
Brief Title: The Feasible Research of Infrared Endoscope to Diagnose Early Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Shuhui Liang, Associated Professor, Xijing Hospital of Digestive Diseases
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRI-EGC
Record Dates: First submitted 2016-02-29; First posted 2016-03-17 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Early Gastric Cancer
Keywords: Early gastric cancer; Infrared endoscope
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cancer group (Experimental): All patients receive the infrared endoscopy after injecting indocyanine green（ICG） intravenously.
  Interventions: Device: infrared endoscopy
- Non-cancer group (Other): All patients receive the infrared endoscopy after injecting ICG intravenously.
  Interventions: Device: infrared endoscopy

INTERVENTIONS:
Device: infrared endoscopy — Firstly use standard white light and narrow-band imaging to observe the lesion, and then inject the contrast medium ICG, after 2 minutes,switch to infrared light to observe, record the image data, then accomplish the examination.

SUMMARY:
The gastric cancer is the second most frequently diagnosed cancer and the third leading cause of cancer death in China.80%-90% patients were detected at middle and later stage.The five-year survival rate for advanced gastric cancer patients is less than 10% due to the shortage of effective treatment method.The five-year survival rate for early gastric cancer patients is beyond 90%.The reason for poor diagnosis and treatment is that current methods do not achieve the diagnosis of early gastric cancer.Endoscopy with biopsy is still the main method for confirming gastric cancer.But it is limited to identify early gastric cancer and it leads to the low diagnostic rate of early gastric cancer.

Infrared endoscopic imaging is a new great potential method of diagnosis of early gastric cancer, since the first report in the 1990s, people have been exploring in this field. Through intravenous injection of exogenous contrast medium, such as the indocyanine green, it makes mucosal lesions highlight,and avoids the interference of background light.If specific target molecular is linked to the contrast medium,the specific imaging of the lesion can be presented. What is more,due to the strong penetration power of infrared light,its imaging depth also increases significantly.Indocyanine green had also been demonstrated safe in clinical studies and widely used. On this basis,we apply for the research about near-infrared endoscopy to diagnose early gastric cancer,and discuss its feasibility of the infrared endoscopy to diagnose early gastric cancer and clinical value.

DETAILED DESCRIPTION:
The gastric cancer is the second most frequently diagnosed cancer and the third leading cause of cancer death in China.80%-90% patients were detected at middle and later stage.The five-year survival rate for advanced gastric cancer patients is less than 10% due to the shortage of effective treatment method.The five-year survival rate for early gastric cancer patients is beyond 90%.The reason for poor diagnosis and treatment is that current methods do not achieve the diagnosis of early gastric cancer.Endoscopy with biopsy is still the main method for confirming gastric cancer.But it is limited to identify early gastric cancer and it leads to the low diagnostic rate of early gastric cancer.

Accurate diagnosis for early gastric cancer and the pretherapeutic estimation of the invasion depth is desired to determine suitable treatment.Presently,endoscopic submucosal dissection is the new effective minimally invasive treatment for early gastric cancer,which preserve the entire stomach and improve the patient's postoperative quality of life.But the estimation of invasion depth of gastric cancers should be confirmed before operation.

Recently,some research suggest that narrow banding imaging and endoscopy ultrasonography are considered established means of diagnosis for early gastric cancer and depth.No formal quantitative review of the available evidence has been published that narrow banding imaging or endoscopy ultrasonography could accurately diagnose early gastric cancer and evaluate the invasive depth.This means still has great limitations.The sensitivity of narrow banding imaging diagnosis is only 60% which its high false positive rate,shorter wavelength and lighter penetration,and the result is influenced by histologic variety of early gastric cancer and inflammatory changes in the background mucosa;Although endoscopy ultrasonography achieves a diagnostic accuracy of over 80%,and its tomographic views facilitate objective assessments,it is occasionally difficult to obtain images with adequate quality, and its evaluation is highly dependent on operators' proficiency levels.

Infrared endoscopic imaging is a new great potential method of diagnosis of early gastric cancer, since the first report in the 1990 s, people have been exploring in this field. Through intravenous injection of exogenous contrast medium, such as the indocyanine green, it makes mucosal lesions highlight,and avoids the interference of background light.If specific target molecular is linked to the contrast medium,the specific imaging of the lesion can be presented. What is more,due to the strong penetration power of infrared light,its imaging depth also increases significantly.Indocyanine green had also been demonstrated safe in clinical studies and widely used, such assessment of liver function tests.

At present,the research in this aspect is very few, a few clinical research results show that infrared endoscopic imaging has a larger value for differentiating between early gastric cancer and gastric adenoma, and the difference between early gastric cancer and gastric lesions is significantly correlated with the depth of cancer invasion.

However, there is not a system research about the infrared imaging characteristics of gastric cancer and different precancerous status,and there is no infrared endoscopic imaging assessment criteria for diagnosis of gastric cancer.

Recently, the investigators have completed the experiments on animals about infrared imaging, the results prove that it has good specificity to identify tumor lesion. On this basis,the investigators apply for the research about near-infrared endoscopy to diagnose early gastric cancer,and discuss its feasibility of the infrared endoscopy to diagnose early gastric cancer and clinical value.

ELIGIBILITY:
Inclusion Criteria:

1. Age：18-70
2. Sex：unlimited；
3. Group 1：patients with EGC，willing to receive treatment under endoscopy（EMR/ESD）
4. Group 2：patients for screening，or have some general symptoms dyspepsia、epigastric pain）who need to be examined by endoscopy
5. Informed consent issued

Exclusion Criteria:

1. Severe liver and kidney disease;
2. Iodine, seafood or other severe allergies history；
3. Patients with severe heart or pulmonary disease which is not suitable for endoscopic examination
4. Higher blood risk of esophageal varices
5. Pregnant or lactating female
6. Without patient's consent
7. The investigator considers other condition which is not suitable for participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-06 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
the lesion of early gastric cancer by infrared endoscopy | up to two years
  confirming that the lesion of early gastric cancer can gather indocyanine green and can be observed by the infrared endoscopy.

SECONDARY OUTCOMES:
the invasive depth of early gastric cancer by infrared endoscopy | two years

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, M.D., Prof., Study Director — Xijing Hospital of Digestive Diseases
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes